CLINICAL TRIAL: NCT07384390
Title: An Open-Label, Dose-Escalation, Multiple Administration, Exploratory Clinical Study to Evaluate the Safety, Tolerability, and Anti-tumor Activity of TH-CART-027 Cell Injection in Subjects With Recurrent or Progressive Grade 4 Glioma
Brief Title: TH-CAR-027 for Grade 4 Gliomas
Status: Not yet recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Shanghai Tongji Hospital, Tongji University School of Medicine (Other)
Responsible Party: Principal Investigator, Chun Luo, Director， Prof., Shanghai Tongji Hospital, Tongji University School of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2025IIT-C0019
Record Dates: First submitted 2026-01-26; First posted 2026-02-03 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-02

CONDITIONS: R/R Grade 4 Glioma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TH-CART-027 (Experimental): mutliple-dosing, intratumoral and/or intraventricular infusion
  Interventions: Drug: TH-CART-027

INTERVENTIONS:
Drug: TH-CART-027 — Multiple-dosing, intratumoral and/or intraventricular infusion

SUMMARY:
This is an open-Label, dose-escalation, multiple administration, exploratory clinical study to evaluate the safety, tolerability, and anti-tumor activity of TH-CART-027 cell injection in subjects with recurrent or progressive grade 4 glioma

ELIGIBILITY:
Inclusion Criteria:

* 1. Voluntarily participate in the clinical trial; fully understand and are informed about this study and sign the informed consent form; willing and able to comply with and complete all trial procedures.

  2. Male or female patients aged ≥18 years and ≤75 years. 3. Disease Status: Diagnosis of Grade 4 glioma as defined by the 2021 WHO Classification of Tumors of the Central Nervous System, including but not limited to glioblastoma, Grade 4 astrocytoma, and diffuse hemispheric glioma. Subjects must have experienced relapse or progression following standard therapy and are unsuitable for or refuse further surgical resection. Subjects with specific genetic mutations (e.g., NTRK gene fusion or BRAF V600E mutation) must have progressed after receiving corresponding targeted therapy to be eligible. Documentation of relapse/progression must include imaging (MRI or PET) or histopathological confirmation.

  4. B7-H3 Expression: ≥30% positivity for B7-H3 molecule in primary/relapsed tumor tissue by pathological testing. B7-H3 positivity is defined as: the percentage of B7-H3-positive tumor cells among total viable tumor cells in non-necrotic tumor tissue areas ≥30%.

  5. Karnofsky Performance Status (KPS) score ≥60, or Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.

  6. Adequate venous access for peripheral blood mononuclear cell (PBMC) collection.

  7. Left ventricular ejection fraction (LVEF) ≥40% by cardiac ultrasound within one month prior to screening.

  8. Resting oxygen saturation ≥95% while breathing room air. 9. Laboratory tests must meet the following criteria within the specified timeframe prior to screening:
  1. Hematological Function: Absolute neutrophil count (ANC)≥1.5×10^9/L, hemoglobin ≥90 g/L, platelet count≥100×10^9/L, absolute lymphocyte count≥0.15×10^9/L. No transfusion,granulocyte (macrophage)colony-stimulating factor, recombinant human erythropoietin, recombinant human thrombopoietin, thrombopoietin receptor agonist, recombinant human interleukin-11, or other supportive therapy within 14 days prior to the test.
  2. Liver Function: Total bilirubin≤1.5×upper limit of normal (ULN) (except for patients with Gilbert's syndrome characterized by persistent or recurrent unconjugated hyperbilirubinemia in the absence of hemolysis or hepatic pathology); Alanine aminotransferase (ALT) and Aspartate aminotransferase (AST)≤2.5×ULN.
  3. Renal Function: Serum creatinine ≤1.5×ULN.
  4. Coagulation: Prothrombin time (PT) or activated partial thromboplastin time (aPTT) or international normalized ratio (INR) ≤1.5 ×ULN, in the absence of therapeutic anticoagulation.

     10. Female subjects of childbearing potential must have a negative urine or serum pregnancy test. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test is required. Female subjects of childbearing potential must use highly effective contraception from the start of the trial until 6 months after the last dose of study treatment. Sexually active males, who have not undergone vasectomy, must agree to use barrier contraception from the start of the trial until 6 months after the last dose of study treatment.

     Exclusion Criteria:

     Subjects with a known history of severe allergy to any component of the investigational product.

     Pregnant or lactating women. Body weight <40 kg.

     Viral Infections:

  <!-- -->

  1. Seropositivity for HIV antibody or positive serological test for Treponema pallidum (syphilis).
  2. Hepatitis B surface antigen (HBsAg) positivity with peripheral blood HBV DNA levels above the upper limit of normal.
  3. Hepatitis C virus (HCV) antibody positivity with detectable peripheral blood HCV RNA.

     Medical History and Concurrent Conditions:

  <!-- -->

  1. Having undergone carmustine wafer implantation surgery within the past 6 months.
  2. Known or suspected active autoimmune diseases, including but not limited to Crohn's disease, rheumatoid arthritis, systemic lupus erythematosus, etc.
  3. Current requirement for systemic immunosuppressive therapy or, in the investigator's judgment, a need for long-term immunosuppressant use during the study period. Intermittent use of topical, inhaled, or intranasal corticosteroids is allowed.
  4. Uncontrolled psychiatric disorders. Or subjects with a medical or psychiatric history that, in the investigator's opinion, could increase the risk associated with study participation or administration of the study drug, or could interfere with the interpretation of results.
  5. Toxicities from prior anticancer therapy have not recovered to ≤ Grade 1 per CTCAE version 5.0 (except for alopecia and other events deemed tolerable by the investigator).
  6. Participation in another interventional clinical trial within the past 1 month.
  7. Prior treatment with any CAR-T therapy or other gene therapy.
  8. Any severe or poorly controlled medical condition that, in the investigator's opinion, may increase the risk associated with study participation or study drug administration, or impair the subject's ability to receive the investigational product. This includes, but is not limited to, cardiovascular/cerebrovascular diseases, renal insufficiency, pulmonary embolism, coagulopathy or requirement for long-term anticoagulation therapy, active or uncontrolled infection requiring systemic treatment.
  9. History or presence of other malignancies within the past 3 years, except for adequately treated non-melanoma skin cancer or carcinoma in situ (e.g., cervical, bladder, breast).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-01-30 (Estimated); Primary Completion 2028-08-31 (Estimated); Study Completion 2029-08-31 (Estimated)

PRIMARY OUTCOMES:
Safety：Incidence of Dose Limiting Toxicity (DLT) | 28 days after the first TH-CART-027 infusion
  Limiting toxicity type, incidence, and severity of dose limiting toxicities (DLTs) within 28 days after the first TH-CART-027 infusion
Safety：Incidence and severity of adverse events (AEs) | Six months post CAR-T cells infusion.
  To evaluate possible adverse events after TH-CAPT-027 infusion, including the incidence and severity of AEs.

SECONDARY OUTCOMES:
Overall survival (OS) | 12 and 24 months post CAR-T cells infusion
  Time from treatment initiation to death from any cause.
Objective response rate (ORR) | 3 months post CAR-T cells infusion
  The assessment will be based on the investigator's evaluation of imaging evaluations, with efficacy evaluated according to the Response Evaluation Criteria in Solid Tumors (RECIST 1.1). ORR refers to the proportion of patients with objective evidence of achieving a Complete Response (CR) or Partial Response (PR). Where applicable, responses recorded after disease progression or initiation of non-investigational anticancer therapy will be excluded
Progression Free Survival (PFS) | 1 year post CAR-T cells infusion
  Defined as the time from initiation of the investigational drug to the first occurrence of progressive disease (PD) or death from any cause in the absence of documented PD. If no tumor progression is observed and the subject does not die during the study period, the analysis cutoff date will be determined as the date of the last tumor assessment
Disease Control Rate (DCR) | 1 year post CAR-T cells infusion
  Defined as the proportion of patients achieving Partial Response (PR), Complete Response (CR), or Stable Disease (SD) according to RECIST 1.1 criteria, relative to the total number of cases in the study

IPD SHARING:
Plan to Share IPD: No